CLINICAL TRIAL: NCT06968819
Title: The Effect of a Virtual Reality-Based Robot-Assisted Dual-Task Intervention on Motor Rehabilitation and Psychological Distress in Patients With Inflammatory Myopathy: a Randomised Controlled Trial
Brief Title: Virtual Reality and Robotics in Inflammatory Myopathy Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Geriatrics, Rheumatology and Rehabilitation, Poland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: nigrr_myopathy
Record Dates: First submitted 2025-04-18; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Inflammatory Myopathy
Keywords: virtual reality; robot assisted rehabilitation; dual-task intervention; randomised controlled trial
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-immersive virtual reality based rehabilitation (Experimental)
  Interventions: Other: Non-immersive virtual reality
- Standard physical therapy (Active Comparator)
  Interventions: Other: Standard physical therapy

INTERVENTIONS:
Other: Non-immersive virtual reality — Non-immersive virtual reality-based robot-assisted intervention includes balance and coordination training, muscle strengthening exercises as well as cognitive stimulation activities on an interactive treadmill, stabilometric platform and robot-assisted upper limb rehabilitation device. In addition, the experimental group takes part in group sessions featuring active and isometric exercises or motor coordination training.
  Arms: Non-immersive virtual reality based rehabilitation
Other: Standard physical therapy — Participants receive standard physical therapy, which includes individual sessions focused on muscle strengthening, balance training, stretching, suspension therapy, and treadmill exercises. In addition, they take part in group sessions featuring active, isometric exercises or motor coordination training.
  Arms: Standard physical therapy

SUMMARY:
The goal of this clinical trial is to learn if a virtual reality based robot assisted dual task intervention leads to better rehabilitation effects than standard physical therapy in patients with inflammatory myopathy. The main question it aims to answer is whether a non-immersive virtual reality based rehabilitation improves muscular strength and relieves psychological distress to a greater extent than standard physical therapy conducted by physiotherapists.

* Participants will be divided into intervention and control group.
* The control group will participate in a standard rehabilitation program consisting of exercise sessions with physiotherapists.
* The intervention group will train on the robotic devices (Zebris treadmill, Alfa stabilometric platform, Diego robotic set).
* Both group will train from 4 to 6 weeks, 5 times a week.
* 6 weeks after completing the rehabilitation program, patients will return for a follow-up assessement.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 y.o,
* meeting the Bohan/Peter criteria for myositis or the ENMC criteria for immune-mediated necrotising myopathy and for inclusion body myositis,
* reduced muscular strength defined by ≤ 64/80 result in MMT-8 and/or ≤ 7/10 result in MMT in ≥ 1 proximal muscle group

Exclusion Criteria:

* severe cardiopulmonary diseases,
* concurrent malignancies,
* severe psychiatric disorders
* injuries and comorbidities preventing exercise participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | change from baseline at week 4-6 and week 10-12
  The Manual Muscle Testing (MMT-8) evaluates the strength of eight designated muscle groups: Deltoid, Biceps, Wrist extensors, Quadriceps, Ankle dorsiflexors, Neck flexors, Gluteus medius, and Gluteus maximus. Each muscle group is rated on a scale from 0 to 10 points, with the total score ranging from 0 to 150.
Muscle endurance | change from baseline at week 4-6 and week 10-12
  The Functional Index-3 (FI-3) involves the assessment of the number of repetitions of shoulder flexion, neck flexion, and hip flexion. Maximum number of repetitions for shoulder flexion and hip flexion is 60 each. Maximum number of repetitions for neck flexion is 30. The total score (summation of the individual tasks divided by 3) ranges from 0 to 50.

SECONDARY OUTCOMES:
Functional exercise capacity and aerobic fitness | change from baseline at week 4-6 and week 10-12
  Ergospirometry assesses maximal oxygen uptake (VO₂max), defined as the maximum amount of oxygen consumed per minute per kilogram of body weight (mL/kg/min). A higher VO₂max reflects greater aerobic fitness and functional exercise capacity.
Health Assessment Questionnaire | change from baseline at week 4-6 and week 10-12
  Self-assessment tool to measure the functional status. The score ranges from 0 to 3, where 0 indicates no difficulty in performing daily physical activities, and 3 indicates an inability to perform them
Gait analysis | change from baseline at week 4-6 and week 10-12
  Gait analysis is performed on a force-sensing Zebris® treadmill. Step length, stride length, cadence, velocity, step time, stride time, single limb support are measured.
Stance analysis | change from baseline at week 4-6 and week 10-12
  Centre of pressure path length measured with the use of Zebris® treadmill system
Functional exercise capacity | change from baseline at week 4-6 and week 10-12
  In a Six Minute Walk Test (6MWT) a total distance walked by a patient (in meters) is recorded. A greater distance covered indicates better physical performance and higher functional capacity.
Serum activity of creatine phosphokinase | change from baseline at week 4-6 and week 10-12
  Reference range: 39-308 U/L
Serum activity of lactate dehydrogenase | change from baseline at week 4-6 and week 10-12
  Reference rage: 135-225 U/L
Serum activity of C reactive protein | change from baseline at week 4-6 and week 10-12
  Reference range: < 5 mg/L
Patient Global Activity | change from baseline at week 4-6 and week 10-12
  self-assessment tool to measure patient's overall disease activity using a 10 cm visual analogue scale where 0 cm indicates no evidence of disease activity and 10 cm indicates extremely active or severe disease activity
Self-reported quality of life | change from baseline at week 4-6 and week 10-12
  The WHOQOL-BREF questionnaire is used for self-assessment across four domains: physical health, psychological health, social relationships, and environment. Each item is scored from 1 (very unhappy) to 5 (very happy). Total score ranges from 0 to 100.
Depression, Anxiety, Stress | change from baseline at week 4-6 and week 10-12
  DASS-42 (depression, anxiety, stress scale). The score in each category (depression, anxiety, stress) ranges from 0 to 42. A higher score is an indicator of greater intensity of the assessed trait.
Fatigue | change from baseline at week 4-6 and week 10-12
  Modified Fatigue Impact Scale (MFIS): the score ranges from 0 to 84, where 0 indicates the lowest level of fatigue and 84 indicates the highest level of fatigue
Pain coping strategies | change from baseline at week 4-6 and week 10-12
  Pain coping strategies questionnaire (CSQ), the score in each strategy (distraction, re-evaluation of pain, catastrophizing, ignoring sensations, praying/hoping, declaring coping, increased behavioral activity) ranges from 0 to 6. The higher the score, the greater the importance attributed to the given coping strategy for pain.
Personality domains | baseline
  Big Five Inventory questionnaire (BFI-2) is used to assess 5 personality domains: extraversion, agreeableness, conscientiousness, neuroticism and openness. Each statement is rated from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate a greater tendency toward that personality trait.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Markowska, Principal Investigator — National Institute of Geriatrics, Rheumatology and Rehabilitation; Beata Tarnacka, Professor, Principal Investigator — National Institute of Geriatrics, Rheumatology and Rehabilitation; Justyna Frasuńska, PhD, Principal Investigator — National Institute of Geriatrics, Rheumatology and Rehabilitation
Locations (1):
- National Institute of Geriatrics, Rheumatology and Rehabilitation, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No